CLINICAL TRIAL: NCT06969092
Title: A Study on the Correlation Between Oral Health and Delirium in Surgical Inpatients
Status: Recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-25-004
Record Dates: First submitted 2025-04-26; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Oral Health
Keywords: Oral Health; Oral Frailty; Surgical; Surgery; Delirium; Endotracheal Intubation; Cognitive Function
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Oral Frailty Group
  Interventions: Other: Oral Frailty
- Non-Oral Frailty Group

INTERVENTIONS:
Other: Oral Frailty — The exposure factor is the presence of oral frailty in patients before surgery, and oral frailty is evaluated using a scale.
  Groups: Oral Frailty Group

SUMMARY:
Delirium is a clinical syndrome characterized by acute attention deficits, altered consciousness, and fluctuating cognitive dysfunction, typically triggered by multifactorial causes such as physical illness, medication use, or postoperative stress . As the most common complication in hospitalized patients, delirium is highly prevalent among elderly surgical populations, with postoperative delirium (POD) occurring in 7.5%-27.5% of cases, and rates rising to 50%-70% in intensive care unit (ICU) patients . Its onset is closely associated with poor prognoses, including long-term postoperative cognitive decline , increased mortality, prolonged hospitalization, and elevated healthcare costs (annual costs in the United States ranging from 38billionto152 billion) . Early prevention and screening of POD are therefore critical to improving patient outcomes and reducing healthcare burdens.

Surgical patients' oral health issues exhibit multifactorial pathogenesis: intrinsic factors (e.g., age-related tooth loss, malnutrition-induced mucosal repair impairment, and chewing dysfunction due to reduced skeletal muscle mass) and iatrogenic factors (e.g., endotracheal intubation trauma, salivary secretion suppression from analgesics, and inadequate perioperative oral care). Poor oral health in hospitalized patients is often attributable to aging, physical dependence, cognitive decline, malnutrition, low skeletal muscle mass/strength, and comorbidities. The recently proposed concept of "Oral Frailty"-a progressive decline in oral structure and function-strongly predicts physical frailty, dysphagia, malnutrition, long-term care needs, and mortality in community-dwelling older adults

The impact of oral health on cognitive function may involve three pathways :

Mechanical pathway: Tooth loss disrupts masticatory motor function, reduces cerebral blood flow, and diminishes afferent stimulation from peripheral receptors (e.g., periodontal ligaments), leading to weakened neural connectivity and regional brain atrophy.

Neurodegenerative pathway: Tooth loss accelerates neuronal damage via apoptosis and mitophagy, increasing amyloid-beta deposition in the brain.

Inflammatory/metabolic pathway: Systemic inflammation, metabolic dysregulation, microbial-gut-brain axis interactions, and activation of microglia/astrocytes drive neuroinflammatory cascades in the central nervous system.

Given these connections, oral frailty may act as an independent risk factor distinct from general frailty and a potential contributor to POD. These findings suggest that oral frailty could serve as a unique biomarker for perioperative neurocognitive disorders, mediating their pathogenesis. Systematic investigation into the spatiotemporal relationship and mechanisms linking oral health to POD in surgical patients holds significant clinical value for developing multimodal prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years scheduled for elective cardiac or thoracic surgery requiring endotracheal intubation.

Patients without consciousness impairment, able to cooperate with the investigation.

Patients or their legal guardians informed about the study's purpose, methodology, and content, with signed informed consent forms.

Exclusion Criteria:

* Patients with pre-existing oral conditions (e.g., xerostomia, oral mucosal lesions) prior to mechanical ventilation.

Patients with a history of radiotherapy, chemotherapy, or corticosteroid use before surgery.

Patients experiencing intraoperative mortality.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective cardiac surgery under general anesthesia requiring endotracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Delirium | Within One Week Postoperatively
  First, assess the patient's consciousness using the Richmond Agitation-Sedation Scale (RASS). This scale categorizes sedation levels into 10 grades, ranging from +4 (combative) to -5 (comatose), with each score corresponding to a distinct state of consciousness. Next, perform delirium assessment using the Confusion Assessment Method for the ICU (CAM-ICU).he Chinese version of CAM-ICU evaluates delirium through four domains:
  * fluctuating Mental Status ②Attention Deficits
    * Disorganized Thinking ④Altered Consciousness Clarity A delirium diagnosis is confirmed if criteria ① and ② are met, along with either ③ and/or ④.
  Consciousness comprises two components: arousal level and awareness content. To assess delirium, begin by evaluating arousal level using the RASS. If the patient's RASS score is not -4 or -5 (indicating adequate arousal), proceed with delirium evaluation.

SECONDARY OUTCOMES:
dysphagia | 48 hours after removal of the endotracheal tube
  The Kubota Water Swallowing Test is used to evaluate a patient's swallowing function and is a classic bedside assessment method. The evaluation criteria are as follows:
  The patient sits upright and drinks 30 mL of warm water. Observe the time required and presence of coughing during swallowing.
  Grading and Criteria:
  Grade 1 (Excellent): Swallows all 30 mL smoothly in one attempt without coughing.
  Grade 2 (Good): Swallows in two or more attempts without coughing.
  Grade 3 (Fair): Swallows in one attempt but with coughing.
  Grade 4 (Poor): Swallows in two or more attempts with coughing.
  Grade 5 (Very Poor): Frequent coughing, unable to swallow completely.
  Interpretation of Swallowing Function:
  Normal: Grade 1, completed within 5 seconds.
  Suspicious: Grade 1 with completion time exceeding 5 seconds or Grade 2.
  Abnormal: Grades 3-5.
appetite | 48 hours after removal of the endotracheal tube
  The Simplified Nutritional Appetite Questionnaire (SNAQ) is used to assess patients' appetite. It evaluates nutritional status by inquiring about appetite, food intake volume, perception of food taste, and related factors. For predicting the risk of 5% and 10% weight loss, the SNAQ demonstrates sensitivity and specificity of 81.3% and 76.4% (for 5%) and 88.2% and 83.5% (for 10%), respectively. The questionnaire comprises 6 items, each scored on a 1-5 point Likert scale. A total score <14 indicates a high-risk patient for weight loss, likely classified as an anorexic individual requiring intervention.
Serum albumin | Postoperative serum albumin levels are routinely assessed within the first week after surgery.
  Serum albumin is a mandatory laboratory test for postoperative patients, measured via blood sampling.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xinhua hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No